CLINICAL TRIAL: NCT03691883
Title: Design of an Integrative Algorithm for Staging Tuberculosis to Improve Clinical Management.
Brief Title: Design of an Integrative Algorithm for Staging Tuberculosis
Acronym: STAGE-TB
Status: Recruiting | Type: Observational
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Hospital Universitari Vall d'Hebron (Drassanes) (Unknown); Servicios Clínicos de Barcelona (Unknown); Germans Trias i Pujol Hospital (Other); Hospital Sant Joan de Deu (Other); Hospital del Mar (Other)
Responsible Party: Sponsor
Other Study IDs: STAGE-TB
Record Dates: First submitted 2017-09-03; First posted 2018-10-02 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Tuberculosis
Keywords: tuberculosis, infectious diseases
MeSH Terms: conditions — Tuberculosis; Communicable Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples With DNA — Bloood samples for determination of DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- TB patients: TB patients diagnosed and followed-up in Barcelona, at the following Hospitals/Clinics: Servicios Clínicos, Hospital Universitari Germans Trias i Pujol, Hospital Universitari Vall d'Hebron-Drassanes, Hospital del Mar.

SUMMARY:
Tuberculosis is a chronic infectious disease that affects 10 million people, 300 in the city of Barcelona, every year. With serious consequences at public health level, it is associated with other diseases, and generated and influenced by many social and psychological factors. This study aims to stage tuberculosis disease by an integrative approach.

DETAILED DESCRIPTION:
Tuberculosis is a chronic infectious disease that affects 10 million people, there are 300 new cases 300 in the city of Barcelona, every year. Tuberculosis has serious consequences at public health level. It is associated with other diseases, and generated and influenced by many social and psychological factors. This study aims to stage tuberculosis disease by a novel integrative approach.

ELIGIBILITY:
Inclusion Criteria:

* TB diagnosis (all forms), microbiologically confirmed (by AFB+, GenXpert+ or Culture+)
* Clinical management of the patients being done at Servicios Clínicos, Hospital Universitari Vall d'Hebron-Drassanes or Hospital Universitari Germans Trias i Pujol.

Exclusion Criteria:

* Not consenting to data/samples donation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: TB patients which clinical management is done at the following clinical centers: Servicios Clínicos, Hospital Universitari Vall d'Hebron-Drassanes or Hospital Universitari Germans Trias i Pujol.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Clinical changes | timepoints 0 (at inclusion), at month 2 and month 6 (and month 12 if MDR/XDR)
  Changes in clinical status
Microbiological changes | timepoints 0 (at inclusion), at month 2 and month 6 (and month 12 if MDR/XDR)
  Changes in microbiological cultures

SECONDARY OUTCOMES:
Changes in Biomarkers values | timepoints 0 (at inclusion), at month 2 and month 6 (and month 12 if MDR/XDR)
  Changes in the biomarkers along time assessed by using analyzing parameters in blood and urine samples (by ELISA and LUMINEX)
Radiological Score Value | timepoints 0 (at inclusion), at month 2 and month 6 (and month 12 if MDR/XDR)
  Changes in the BCN-SA Radiological Score Value. This Score assesses the sum of acute and chronic findings in the chest X-ray. Per each finding, a maximum score of 8 is recorded. The total score value is calculated by adding all the individual findings score values. Higher values of total score represent a worse outcome.
Changes in SGRQ score | timepoints 0 (at inclusion), at month 2 and month 6 (and month 12 if MDR/XDR)
  Changes in Health Quality of Life measures along time assessed by using the Saint George's Respiratory Questionnaire (SGRQ, numeric score). It measures 3 subscales (symptoms/activity/impacts) and The Total score is calculated by summing all positive responses in the questionnaire and expressing the result as a percentage of the total weight for the questionnaire. Higher values represent a worse outcome.
Changes in Kessler-10 score | timepoints 0 (at inclusion), at month 2 and month 6 (and month 12 if MDR/XDR)
  Changes in Health Quality of Life measures along time assessed by using the questionnaire Kessler-10 (K10, numeric score). Higher values represent a worse outcome.
Changes in Health Quality of Life measures along time using BCN-Q questionnaire | timepoints 0 (at inclusion), at month 2 and month 6 (and month 12 if MDR/XDR)
  Changes in Health Quality of Life measures along time using BCN-Q questionnaire (descriptive questionnaire).

CONTACTS AND LOCATIONS:
Overall Officials: Cris Vilaplana, MD, PhD, Principal Investigator — Fundació Institut Germans Trias i Pujol
Locations (5):
- Spain (5):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Sant Joan de Déu, Esplugues de Llobregat, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron-Drassanes, Barcelona
  - Servicios Clínicos de Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: Undecided
IPD that underlie results in a publication might be shared with other researchers

REFERENCES:
- [Background] Romero-Tamarit A, Valles X, Munar-Garcia M, Espinosa-Pereiro J, Saborit N, Tortola MT, Stojanovic Z, Roure S, Antuori A, Cardona PJ, Soriano-Arandes A, Martin-Nalda A, Espiau M, de Souza-Galvao ML, Jimenez MA, Noguera-Julian A, Molina I, Casas X, Dominguez-Alvarez M, Jove N, Gogichadze N, L Fonseca K, Arias L, Millet JP, Sanchez-Montalva A, Vilaplana C. A longitudinal prospective study of active tuberculosis in a Western Europe setting: insights and findings. Infection. 2024 Apr;52(2):611-623. doi: 10.1007/s15010-024-02184-2. Epub 2024 Feb 13. PMID 38349459
- [Background] Roure S, Valles X, Sopena N, Benitez RM, Reynaga EA, Bracke C, Loste C, Mateu L, Antuori A, Baena T, Portela G, Llussa J, Flamarich C, Soldevila L, Tenesa M, Perez R, Plasencia E, Bechini J, Pedro-Botet ML, Clotet B, Vilaplana C. Disseminated tuberculosis and diagnosis delay during the COVID-19 era in a Western European country: a case series analysis. Front Public Health. 2023 May 18;11:1175482. doi: 10.3389/fpubh.2023.1175482. eCollection 2023. PMID 37275492
- [Result] Pujol-Cruells A, Vilaplana C. Specific Interventions for Implementing a Patient-Centered Approach to TB Care in Low-Incidence Cities. Front Med (Lausanne). 2019 Nov 26;6:273. doi: 10.3389/fmed.2019.00273. eCollection 2019. PMID 31850353
- See also: Institutional webpage- Experimental TB Unit — https://www.germanstrias.org/en/research/infectious-diseases/2/experimental-tuberculosis-unit-ute